CLINICAL TRIAL: NCT00993733
Title: Assessing the Impact of Two Methods of Continuous Veno-venous Hemodiafiltration on Time Nursing Work in Intensive Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study has never been started
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1008019; 2010-A00695-34 (Other: AFSSAPS)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Acute Renal Failure
Keywords: hemodiafiltration; cost; dialysis solution; acute renal failure; intensive care unit
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CVVHDF on-line (Experimental): CVVHDF using a central water treatment plant, providing dialysate directly to the patient. They will perform a continuous veno-venous haemodiafiltration.
  Interventions: Procedure: Continuous veno-venous haemodiafiltration
- classical CVVHDF (Experimental): CVVHDF using a mobile generator with dialysate bags. They will perform a continuous veno-venous haemodiafiltration.
  Interventions: Procedure: Continuous veno-venous haemodiafiltration

INTERVENTIONS:
Procedure: Continuous veno-venous haemodiafiltration — Dialysis procedure administrated to the patients with acute renal failure
  Other Names: Classical CVVHDF : dialusate generator Prismaflex (HOSPAL); CVVHDF on-line : dialysate generator 5008 (Fresenius)

SUMMARY:
The prevalence of acute renal failure in intensive care is estimated at between 5 and 20% depending on diagnostic criteria retained. And half of patients require the use of hemodialysis. Continuous veno-venous hemodiafiltration (CVVHDF) is one of the hemodialysis technique widely used in intensive care unit.

The CVVHDF is performed at the bedside, by a mobile generator with a semi permeable membrane, a blood circuit, a dialysate circuit and a feedback circuit.

The implementation of a CVVHDF requires the use of large amounts of biological liquid essential to enable the purification of blood during its passage through the artificial kidney.

The objective of this study is to assess time nursing work and the costs of each method.

DETAILED DESCRIPTION:
The prevalence of acute renal failure in intensive care is estimated at between 5 and 20% depending on diagnostic criteria retained. And half of patients require the use of hemodialysis. Continuous veno-venous hemodiafiltration (CVVHDF) is one of the hemodialysis technique widely used in intensive care unit.

The CVVHDF is performed at the bedside, by a mobile generator with a semi permeable membrane, a blood circuit, a dialysate circuit and a feedback circuit.

The implementation of a CVVHDF requires the use of large amounts of biological liquid essential to enable the purification of blood during its passage through the artificial kidney. The biological fluid may be supplied to the generator of CVVHDF in 2 ways:

* The conventional method, the most used: the generator operates with pockets containing dialysis fluid, these pockets to be changed regularly by nurses
* The on-line method: the generator operates with a specific water system supplying the dialysis fluid available in every room of the unit The objective of this study is to assess time nursing work and the costs of each method.

For this, 15 patients will be included in this study. Each patient performs 12 hours of each method (conventional and online), whose order will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated with or beneficiary of a social security category
* Patient with a renal failure requiring a CVVHDF for at least 2 cycles of 12 hours

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
time of nursing work required to realised a CVVHDF as a conventional and on line methods modality of supply compared to a method on-line | Day 1
  The end of the study for the patient corresponds to the end of CVVHDF conventional and on line.

SECONDARY OUTCOMES:
costs of CVVHDF performed using a conventional and on-line methods | Day 1
  The end of the study for the patient corresponds to the end of CVVHDF conventional and on line.

CONTACTS AND LOCATIONS:
Overall Officials: Manolie Mehdi, MD, Principal Investigator — CHU SAINT-ETIENNE

IPD SHARING:
Plan to Share IPD: No